CLINICAL TRIAL: NCT02965339
Title: Evaluation of the Association Between Pre-existing Endothelial Dysfunction and the Onset of Vasoplegia During Cardiac Surgery With Cardiopulmonary Bypass
Acronym: DYVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-05 (PI2015-05)
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Vasoplegia; Endothelial Dysfunction
Keywords: Vasoplegia; endothelial dysfunction; extracorporeal circulation; cardiac surgery
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac surgery patients have many risk factors for endothelial dysfunction (hypertension, atherosclerosis, dyslipidemia, chronic renal failure ...).

It is likely that a significant number of patients suffering from a preexisting endothelial dysfunction. This endothelial dysfunction can be assessed by a molecular approach (determination of NO, ICAM1, VCAM1, IL8, endothelial microparticles ...). Extracorporeal circulation with ischemia-reperfusion causes a breach of particularly important glycocalyx as ischemia-reperfusion injury is. No studies have evaluated the time course of the infringement, and its association with the immediate post-operative complications (SIRS, coagulopathy, vasoplegic syndrome, renal failure). Only one study has regained an association between endothelial dysfunction during cardiac bypass surgery and postoperative cardiac surgery vasoplegic syndrome. A study in noncardiac surgery has regained an association between endothelial dysfunction (assessed by a vasoplegia test) and postoperative acute renal failure. Thus there is some data in the literature to suggest that the occurrence of postoperative complications (SIRS, coagulopathy, capillary leak syndrome, acute circulatory failure vasoplegic and acute renal failure) may result from the interaction between a pre-existing endothelial dysfunction and "operative" aggression (extracorporeal circulation). The onset of complications result from an interaction that depends on the importance of endothelial dysfunction at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years.
* Patient operated on for cardiac surgical myocardial revascularization (CABG) or surgical correction of aortic valve.
* Consent signed.

Exclusion Criteria:

* Standing arrhythmia.
* Pregnant woman.
* curative anticoagulation (warfarin, NANCO, heparin).
* Patient under guardianship.
* Patient Refused to participate.
* Cardiac surgery without CPB.
* bicuspid aortic valve.
* Participation in another study.
* preoperative sepsis.
* Minor or major, under guardianship or trusteeship (art L1121-5, L1121-8 and L1122 1-2)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years, operated on for cardiac surgical myocardial revascularization (CABG) or surgical correction of aortic valve.
  Consent signed.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was the occurrence of vasoplegic syndrome | 6 months
  The primary endpoint was the occurrence of vasoplegic syndrome correlate with markers of endothelial function following: IL8, P-selectin, von Willebrand factor precursor.

SECONDARY OUTCOMES:
Occurrence of vasoplegic syndrome | 6 months
  Occurrence of vasoplegic syndrome correlate with markers of endothelial function following: endothelial microparticles, Von Willebrand factor, VCAM1.
Marker of degradation glycocalyx: | 6 months
  Marker of degradation glycocalyx: syndecan, heparan sulfate.
Inflammatory markers: | 6 months
  Inflammatory markers: leukocytes, CRP, procalcitonin, albumin, TNF alpha, IL-10, IL-6, IL1beta
Markers of blood coagulation | 6 months
  Markers of blood coagulation: Platelet count, PT, APTT, fibrinogen, D dimers, soluble complexes.
Complications | 6 months
  Complications: cardiovascular (vasoplegic syndrome), kidney (KDIGO).
Death | 6 months
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Grégoire GUINOT, Doctor, Principal Investigator — CHU Amiens Picardie
Locations (1):
- CHU De Caen, Caen, France